CLINICAL TRIAL: NCT03756688
Title: Penile Length Restoration in Men With Diabetes Mellitus, Type II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew (Matt) J. Ziegelmann, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-006696
Record Dates: First submitted 2018-11-24; First posted 2018-11-28 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Penile Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Penile Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of four groups:
  1. Penile Traction Therapy (PTT) for 30 min 2x/day x 3 months, followed by no treatment x 3 months
  2. PTT for 30 min 2x/day x 3 months, followed by once weekly (30 minutes) x 3 months
  3. PTT for 30 min 2x/day x 6 months
  4. Control (no treatment)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The provider and outcome assessor will be blinded to the patient's study arm for all length assessments. Additionally, the assessor will be blinded to prior length measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Group 1: Control (No Intervention): No treatment will be administered for the entirety of the study (6 months)
- Group 2: Treatment (Experimental): PTT for 30 min 2x/ day x 3 months, followed by no treatment x 3 months
  Interventions: Device: RestoreX PTT - 3 months
- Group 3: Treatment (Experimental): PTT for 30 min 2x/day x 3 months, followed by once weekly (30 minutes) x 3 months
  Interventions: Device: RestoreX PTT - 6 months
- Group 4: Treatment (Experimental): PTT for 30 min 2x day x 6 months
  Interventions: Device: RestoreX PTT - 6 months

INTERVENTIONS:
Device: RestoreX PTT - 6 months — Penile traction therapy in straight position for all 6 months.
  Arms: Group 3: Treatment; Group 4: Treatment
Device: RestoreX PTT - 3 months — Penile traction therapy in straight position for first phase (3 months)
  Arms: Group 2: Treatment

SUMMARY:
The objective of the current study is to evaluate the efficacy of a novel penile traction device in restoring lost penile length in men with type 2 diabetes.

DETAILED DESCRIPTION:
Men with diabetes mellitus experience sexual dysfunctions at an earlier age and higher rate compared to men without diabetes. One of these sexual dysfunctions includes diminished penile length. It is currently unknown if the decreased length is due to earlier erectile dysfunction or secondary to diabetes itself. Penile traction therapy is one of several treatments which have been used historically to treat decreased penile length, however, to date, no studies have evaluated the role of traction therapy in men with diabetes. To accomplish the study, a population of men from Mayo Clinic with a diagnosis of diabetes, type II will be enrolled and will be randomized to utilize the device for varying amounts of time. Outcomes will be assessed at the 3 and 6 month time points, and the results are to be used with the intent to publish in a scientific journal.

ELIGIBILITY:
Inclusion Criteria:

- Men with Diabetes Mellitus, Type II

Exclusion Criteria:

* Any evidence of end-organ failure attributed to DM (assessed based on medical history / patient history alone)
* Loss of fingers / toes.
* CKD Stage IV or greater.
* Retinopathy
* Myocardial infarction.
* Cerebrovascular accident.
* Indwelling penile prosthesis or prior history of penile prosthesis.
* Peyronie's disease at baseline.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ziegelmann, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Control | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
Started | 28 | 28 | 27 | 27
Completed | 26 | 17 | 19 | 24
Not Completed | 2 | 11 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Control | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment | Total
Number analyzed (Participants) | 28 | 28 | 27 | 27 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (7.0) | 55.1 (5.3) | 55.0 (6.3) | 56.2 (5.4) | 54.9 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 28 | 28 | 27 | 27 | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Penile Length Change Between Baseline and Month 6
Description: Primary objective of this study is to assess penile length pre and post completion of RestoreX traction therapy compared to control groups (no treatment) of Diabetes Type II patients. Measurements were obtained at baseline and 6 months post-prostatectomy.
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: Median change from baseline (cm)
Arm/Group | Group 1: Control | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
Number analyzed (Participants) | 23 | 17 | 18 | 17
Median change from baseline (cm) | 0 [-0.5 to 0.5] | 0.5 [-0.3 to 0.9] | 0.5 [0 to 1.5] | 0.8 [0 to 1.5]

2. Secondary Outcome: Patient Compliance With Traction Therapy
Description: Records of use from daily journals
Time Frame: 6 months
Population: No patients were analyzed in the control arm since the outcome measure was assessing compliance with traction therapy (not administered to controls).
Measure: Mean (Standard Deviation); unit: Percent compliance
Arm/Group | Group 1: Control | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
Number analyzed (Participants) | 0 | 17 | 17 | 21
Percent compliance |  | 93.5 (9.7) | 91.5 (14.3) | 85.2 (21.1)

3. Secondary Outcome: Patient Reported Satisfaction With Traction Therapy at 6 Months.
Description: Likert scale used to assess self-reported overall satisfaction; 1-10 (10 = maximum satisfaction); higher values signify a better outcome. Satisfaction was assessed at 6 months post-prostatectomy.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
Number analyzed (Participants) | 16 | 18 | 20
score on a scale | 7.5 [4.3 to 9] | 8 [6 to 9] | 8 [6.3 to 8.8]

4. Secondary Outcome: Number of Participants With Adverse Events With Use of RestoreX
Description: Adverse events were assessed at 3- and 6-months post-prostatectomy, with results summed and reported as a total.
Time Frame: 3 and 6 months post-prostatectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
Number analyzed (Participants) | 17 | 18 | 20
Participants
  Temporary penile pain (mild) | 2 | 2 | 2
  Pain in other location (unclear if related) | 1 | 0 | 1
  Temporary erythema / discoloration (mild) | 1 | 1 | 4
  Temporary decreased sensation (mild) | 0 | 0 | 1
  Other (unclear if related) | 0 | 0 | 1
  Temporary bleeding from tape (mild) | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With De-novo Peyronie's Disease Development
Description: Subjective question to determine if the patient has developed any new penile curvature, indentation, deformity, or other findings consistent with Peyronie's Disease during the study period
Time Frame: 6 months
Population: Note that reported events represent subjective reporting of penile curvature.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Control | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
Number analyzed (Participants) | 23 | 16 | 18 | 22
Participants | 1 | 2 | 1 | 1

6. Secondary Outcome: Subjective Comparison of Changes in Penile Length
Description: Subjective questions on patient perceived improvement in length (yes/no, qualitative [large, medium, small, none]); note that some groups add to >100% due to the effects of rounding.
Time Frame: 6 months
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Control | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
Number analyzed (Participants) | 17 | 14 | 16 | 20
Percentage of participants
  Subjective improvement in length (% yes) | 0 | 36 | 63 | 65
  Subjective improvement in length (% unsure) | 0 | 36 | 25 | 25
  Subjective improvement in length (no) | 100 | 29 | 13 | 10
  Subjective improvement (large) | 0 | 0 | 9 | 13
  Subjective improvement (medium) | 0 | 50 | 9 | 44
  Subjective improvement (small) | 0 | 50 | 82 | 38
  Subjective improvement (none) | 100 | 0 | 0 | 6

7. Secondary Outcome: Erectile Function Among Groups - Evaluating Change From Baseline to 6 Months.
Description: Standardized questionnaire assessment of erectile function (International Index of Erectile Function standardized questionnaire, Erectile Function Domain [questions 1-5 and 15]). Higher scores are better. Assessments were obtained at baseline and at 6 months post-prostatectomy with the result reported being 6 months minus baseline. Minimum score for the change since baseline = -29 (i.e. 1 minus 30), maximum score = 29 (i.e. 30 minus 1)
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: Control | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
Number analyzed (Participants) | 25 | 17 | 17 | 20
score on a scale | 0 (3.3) | 1.1 (4.6) | 4.2 (10.4) | 4.3 (9.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 6 month period for each subject receiving penile traction treatment.
Description: The control group (Group 1) did not receive penile traction treatment with the traction device. Therefore, adverse events were not collected for this group.
Arm/Group | Group 2: Treatment | Group 3: Treatment | Group 4: Treatment
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 3/28 | 2/27 | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 2: Treatment (N=28) | Group 3: Treatment (N=27) | Group 4: Treatment (N=27)
Transient penile pain (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Transient penile erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Other pain (non-descript location) (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Transient decreased penile sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Temporary bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Other (unclear if related) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03756688/Prot_SAP_000.pdf